CLINICAL TRIAL: NCT05515549
Title: Value of D-dimer Combined With Other Thrombus Molecular Markers in Risk Assessment of VTE in Hospitalized Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Hong Wang, associate chief nurse, Qianfoshan Hospital
Other Study IDs: Hong Wang
Record Dates: First submitted 2022-08-22; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Venous Thromboembolic Disease
Keywords: D-dimer; Thrombus Molecular Markers; venous thromboembolism risk assessment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Venous thrombosis group: The venous blood of the patients under fasting state was collected, and the level of thrombus molecular markers was detected. Color Doppler ultrasound was used as the "gold standard" to determine whether VTE occurred.
  Interventions: Other: Venous blood was collected from patients under fasting state to detect the level of thrombus molecular markers
- Group without venous thrombosis: The venous blood of the patients under fasting state was collected, and the level of thrombus molecular markers was detected. Color Doppler ultrasound was used as the "gold standard" to determine whether VTE occurred.
  Interventions: Other: Venous blood was collected from patients under fasting state to detect the level of thrombus molecular markers

INTERVENTIONS:
Other: Venous blood was collected from patients under fasting state to detect the level of thrombus molecular markers — The venous blood of the patients in fasting state was collected to detect the level of thrombus molecular markers. Color Doppler ultrasound was used as the "gold standard" to determine whether VTE occurred. According to the color Doppler ultrasound diagnosis results, the patients were divided into VTE group and non VTE group.

SUMMARY:
The occurrence of VTE in hospital is an important cause of unexpected death of inpatients, and has become a serious problem faced by hospital managers and clinical medical staff.Under the target of "Improving the Standard Prevention Rate of Venous Thromboembolism" proposed in the "National Medical Quality and Safety Improvement Goal in 2022", it is urgent to establish a highly sensitive VTE risk assessment and monitoring system.At present, VTE risk assessment scale is used for risk screening and monitoring in combination with D-dimer in clinical practice, but D-dimer has low specificity and poor sensitivity, which makes it impossible to accurately assess the risk of venous thrombosis.Therefore, it is very important to explore highly specific molecular markers of thrombosis for VTE risk assessment.This project will analyze the value of single or combined detection of different thrombus molecular markers in VTE risk assessment, establish the best VTE risk assessment scheme, improve the standardized prevention of VTE, realize the early intervention of VTE, truly achieve early detection, early prevention and early treatment, and effectively reduce the occurrence of VTE.

DETAILED DESCRIPTION:
This project is intended to explore the specificity and reliability of single or combined detection of different thrombus molecular markers in venous thrombosis risk assessment by detecting and analyzing the levels of various thrombus molecular markers in VTE high-risk patients, so as to establish the best evaluation strategy for early identification of VTE high-risk patients, build the hospital VTE early warning management system, guide the clinical to formulate targeted graded intervention measures, and effectively reduce the occurrence of VTE. At the same time, it will provide support for the realization of "improving the standard prevention rate of venous thromboembolism" proposed in the national medical quality and safety improvement goal in 2022 and reducing medical risks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Surgical inpatients
* Patients who were assessed as high-risk by venous thrombosis risk assessment after admission (caprini score ≥5)
* Did not receive anticoagulation or thrombolysis before admission
* Patients without chronic cardiovascular disease, autoimmune disease, malignant tumor and other diseases
* Patients without previous history of venous thrombosis of lower limbs
* The molecular markers of thrombus were detected routinely at admission
* The family members of the patients signed informed consent

Exclusion Criteria:

* Abnormal coagulation function due to blood disease or severe liver and kidney dysfunction
* Patients with major trauma or vegetative survival within 3 months
* Patients with long-term use of anticoagulant drugs, glucocorticoids and hemostatic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2023 to December 2024, 300 surgical patients with high risk of venous thrombosis admitted to the First Affiliated Hospital of Shandong First Medical University were selected as the study subjects
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Whether venous thrombosis occurs | On the 13th day after the patient's admission
  On the 13th day after the patient's admission, color Doppler ultrasound will be performed to determine whether the patient has venous thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: hong wang, Principal Investigator — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No